CLINICAL TRIAL: NCT03709069
Title: Effect of Enteral Albumin on Healing of Superficial Partial Thickness Fresh Flame Burns of Adults
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: King Edward Medical University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: Alb-burn
Record Dates: First submitted 2018-10-05; First posted 2018-10-17 (Actual); Last update posted 2018-10-25 (Actual); Status verified 2018-10

CONDITIONS: Partial-thickness Burn

STUDY DESIGN:
Intervention Model Description: One group receives routine diet while other group receives supplemental albumin along with routine diet
Who Masked: Participant, Care Provider, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Traditional Group (No Intervention): Traditional group receives diet from hospital kitchen quantity of which calculated depending on calorie requirement per kg body weight. This diet is same for all burn patients fulfilling the inclusion criteria of the study and it will be labelled as routine diet.
  Wounds of patients will be managed by closed dressing to be changed on every third day.
- Albumin Group (Experimental): Interventional group receiving enteral supplemental albumin 2mg per kg body weight along with routine hospital kitchen diet same as group A and same wound management with closed dressing to be changed on every third day similar to group A.
  Interventions: Dietary Supplement: Albumin supplementation

INTERVENTIONS:
Dietary Supplement: Albumin supplementation — Enteral supplementation by albumin of boiled egg as 2mg per kg body weight.
  Arms: Albumin Group

SUMMARY:
Patients with 10 to 20% Superficial partial thickness fresh flame burn will be recruited. Burn thickness will be confirmed by using Laser Doppler. After randomly allocating into two groups, one group will receive enteral supplemental albumin in the form of boiled egg along with routine diet while other group will receive only routine diet.

Effect of burn healing will be noted in terms of epithelization, oedema, pain and redness and days of hospital stay

DETAILED DESCRIPTION:
Burn is an insult to the living tissues typically skin leading to coagulative necrosis due to extreme of temperature, electricity or chemicals. Burn injuries are a global public health problem with physical, psychological, social and economic implications on patients, their families and society as a whole. According to WHO, about 265,000 people die each year due to burn injuries. Vast majority of burn cases occur in middle and low socioeconomic groups of society. Any age group can be the victim of burn but people belonging to actively working class i.e. young adults (18-40yr) are more susceptible to burn injury. The most common sites of burn occurrence are domestic kitchen and workplaces from upset of receptacles containing hot liquids or directly from flames, electricity or cook stove burst.

Skin has outer covering of epidermis and deeper one is dermis. Burns, from management point of view, can be classified into superficial, superficial partial thickness, deep partial thickness and full thickness depending upon the extent of layers of skin involved. Superficial burns do not need specialized treatment and heal by their own while deep partial thickness and full thickness burns mostly require surgical procedures for management. Patients having superficial partial thickness burn wounds are the group of particular interest in burn centers due to two reasons. Firstly, the majority of burn injuries fall in this group and secondly, these are the wounds which, if managed well, heal in three weeks satisfactorily without any surgical intervention. The superficial partial thickness burn wounds involve damage to epidermis as well as partial dermis and characterized by Slough (yellowish white fibrinous tissue containing proteinacious material, pus and fibrin on wound surface), Erythema (redness of burn skin surface), Ooze (excessive fluid loss).

According to American Burn Association recommendations, patients having superficial partial thickness burn more than 10% body surface area need hospitalization for management. Multiple factors play role in the healing of superficial partial thickness burn wounds like age, co-morbidities (diabetes, HTN, obesity etc), immunosuppressive medications (steroids, chemotherapy) and nutritional status. Management of superficial partial thickness burn wound requires pain management, dressings, topical ointments and culture guided antibiotics. Despite of all these maneuvers, good nutritional support in the form of both micronutrients and macronutrients particularly proteins are critical component of acute burn wound care. Early optimal nutrition administration in management of burn patients particularly involves proteins rich diet due to lot of oozing from large wound surface area, high catabolism of muscles and vast tissue repair.

Protein enrichment of diet, for burn patients, can be achieved by adding albumin, which is easily available from many sources especially egg and plays vital role in burn wound healing. Albumin, synthesized by liver, is one the major proteins which has several important functions. Albumin, composed of essential amino acids, is primary serum binding protein required for transportation of various substances in blood circulation. Albumin administration is much easier through enteral route. Deficit of albumin occurs due to decreased synthesis during inflammatory conditions and, in burns, is further augmented by a shift in distribution of albumin to interstitial space from vascular compartment. A deficiency of albumin level can impair burn wound healing process whereas increased albumin level does not cause significant clinical complication. Hypo-albuminemia caused by wound exudation is the major predictor after injury that results in shock induction secondary to major extracellular fluid loss by increasing vascular permeability.

The rationale of this study is to find out effects of albumin supplementation on hospital stay by affecting healing of superficial partial thickness burn wounds by.

ELIGIBILITY:
Inclusion Criteria:

* 10-20% superficial partial thickness flame burn determined by LASER Doppler.
* Age between 18-40years.
* Fresh burn wound
* Patient with BMI ranging from 18.9-24.9.

Exclusion Criteria:

* Patient not willing to participate
* Any co-morbidities (i.e. DM, HTN, CRF, CCF, CLD)
* Patient with abnormal baseline serum albumin levels
* Patients not taking diet from hospital kitchen
* Patient known allergic to albumin
* Patient put on nil per oral (NPO)

Ages: 18 Years to 40 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 100 (Estimated)
Dates: Start 2018-11-10 (Estimated); Primary Completion 2019-04-09 (Estimated); Study Completion 2019-04-09 (Estimated)

PRIMARY OUTCOMES:
Wound epithelization | 3 weeks
  Wound epithelization will be assessed by photographic image analysis. Serial photographs of wound will be taken on every third day and will be assessed by two independent blinded plastic surgeons to rate for epithelization. The process will be continued till complete epithelization is witnessed.

SECONDARY OUTCOMES:
Effect on pain: PRS | 3 weeks
  Pain will be assessed using Numeral Rating Scale (PRS) by score of 10. Score of 0 will be taken as no pain and score of 10 as maximum pain felt ever by the patient. Pain scoring will be done on every third day till complete healing of wound is acheived.
Change in Oedema | 3 weeks
  Will be assessed clinically as well as by measuring the girth of the area on every third day and change will be recorded

CONTACTS AND LOCATIONS:
Overall Officials: Afzaal Bashir, FCPS,MPhil, Principal Investigator — KEMU Lahore
Locations (1):
- Mayo Burn Center, Lahore, Punjab Province, Pakistan

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Treharne LJ, Kay AR. The initial management of acute burns. J R Army Med Corps. 2001 Jun;147(2):198-205. doi: 10.1136/jramc-147-02-15. PMID 11464415